CLINICAL TRIAL: NCT00128687
Title: Improving Coronary Prevention in a County Health System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Randall Stafford, Professor of Medicine, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 240; R01HL070781 (NIH)
Record Dates: First submitted 2005-08-08; First posted 2005-08-10 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Risk Reduction; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Risk Reduction Behavior; Heart Diseases | interventions — Numbers Needed To Treat

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate Intervention (Experimental): Participants in both arms continue to receive usual medical care throughout the study period. In addition, participants randomized to Immediate Intervention receive intensive case management for Coronary heart disease (CHD) risk reduction for 15 months and then a maintenance program for a minimum of 12 months to assess the durability of initial intervention changes.
  Interventions: Behavioral: risk reduction
- Delayed Intervention (Placebo Comparator): Participants randomized to Delayed Intervention serve as control for Immediate Intervention patients for the first 15 months and then receive intensive case management for 15 months. The switching-over design not only addresses ethical concerns about withholding treatment from half the study sample, but will also enable us to assess whether the intervention had equal impact whether provided to a naïve population or to a group followed in usual care for 15 months.
  Interventions: Behavioral: risk reduction

INTERVENTIONS:
Behavioral: risk reduction — Participants receive intensive case management for CHD risk reduction for 15 months and then a maintenance program for a minimum of 12 months. Lifestyle modification was strongly emphasized as a critical component of achieving CHD prevention goals. Dietary management was emphasized, including recommendation of a low saturated fat (less than 7% of caloric intake), low cholesterol (< 150 mg/day), mainly plant-based diet with calorie restrictions for overweight/obese persons. Stress management and coping skills were emphasized, including a regular exercise regimen (≥ 30 minutes of moderate intensity on most days). Cigarette smokers were encouraged to join a stop smoking program.

SUMMARY:
To examine whether the Stanford Health Education and Risk Reduction Training (HEAR2T) program , a case management approach, can be effectively used to manage the risk of coronary artery disease.

DETAILED DESCRIPTION:
BACKGROUND:

Evidence from extensive population studies and clinical trials shows the effectiveness of risk factor management in reducing morbidity and mortality from coronary artery disease (CAD). These studies have generated important national clinical practice guidelines. Current prevention practices, however, fall short of attaining the goals recommended in these national guidelines. These shortfalls lead to unnecessary CAD disease burden, as well as perpetuation of socioeconomic disparities. Case management proves to augment current CAD prevention activities and improve adherence with national guidelines. The Stanford Health Education and Risk Reduction Training (HEAR2T) program is an innovative, yet well-tested, case management tool which will be evaluated in this study. HEAR2T has been developed and evaluated in several studies at Stanford. It is based upon the social cognitive model of Bandura and uses case managers to work intensely with patients to educate them and change their overall behavior related to health.

DESIGN NARRATIVE:

The Stanford Health Education and Risk Reduction Training (HEAR2T) program will be evaluated in a high-risk population of low socioeconomic status (SES) served by the county health care system of San Mateo County (SMC), California. The study will: 1) enhance the HEAR2T program for use in low-SES populations; 2) implement this program as an integral part of clinical care; 3) implement a randomized controlled trial to evaluate the effectiveness of HEAR2T in lowering aggregate CAD risk; 4) determine if HEAR2T diminishes socioeconomic disparities; 5) estimate HEAR2T's cost effectiveness; and 6) transition the intervention from a research study to an ongoing County CAD case management program. The primary outcome measure will be change in aggregate CAD risk score, calculated from a Framingham model based on individual CAD risk factors. The primary hypothesis is that patients case-management via the HEAR2T model will produce favorable changes in aggregate CAD risk score compared to control patients in usual care. An estimated 200 intervention and 200 usual care patients will be enrolled from four health centers in the SMC system. Usual care patients will crossover to the intervention after 15 months, allowing for additional assessment of the intervention's impact. Continued follow-up of the participants will assess the durability of risk changes achieved during initial intensive case-management. This study will make a critical and innovative contribution to defining optimal disease management in a low-SES population.

ELIGIBILITY:
Abbreviations: FBS = fasting blood sugar, SBP = systolic blood pressure, DBP = diastolic blood pressure, LDL = low-density lipoprotein, HDL = high-density lipoprotein, BMI = body mass index, TC = total cholesterol, TG = triglycerides, HbA1c = hemoglobin A1c.

Inclusion Criteria

* The patient has CAD or CAD risk equivalent (abdominal aortic aneurysm, peripheral vascular disease, transient ischemic attack, stroke, diabetes, or FBS ≥ 126 mg/dL × 2) and has at least one of following: SBP ≥ 130 mmHg, DBP ≥ 80 mmHg, LDL ≥ 100 mg/dL, HDL ≤ 40 mg/dL, TG ≥ 150 mg/dL, FBS ≥ 126 mg/dL, BMI ≥ 30, or is a current smoker.
* The patient does not have CAD or CAD risk equivalent but has at least one of the following: SBP ≥ 160 mmHg, DBP ≥ 100 mmHg, LDL ≥ 190 mg/dL, TC ≥ 240 mg/dL, TG ≥ 500 mg/dL, HbA1c ≥ 8.0%, BMI ≥ 35, or is a current smoker.
* The patient does not have CAD or CAD risk equivalent but has at least two of the following: a) SBP ≥ 140 mmHg or DBP ≤ 90 mmHg, b) HDL ≤ 40 mm/dL or TG ≥ 200 mg/dL, c) LDL ≥ 160 mg/dL or TC ≥ 240 mg/dL, d) FBS ≥ 110 mg/dL × 2, or e) male age ≥ 45 or female age ≥ 55 or with positive family history of CAD.

Exclusion Criteria:

* Resident of long-term facility
* Lack of spoken English or Spanish by patient or household member 18 years or older who can serve as an interpreter
* Moving before end of intervention (30 months)
* Age between 35 and 85 (inclusive)
* Significant comorbidities such as: uncontrolled metabolic disorders (renal failure, liver failure, etc.), active symptoms suggesting acute myocardial infarction or decompensated congestive heart failure, Malignancy or other condition limiting life expectancy, psychiatric disorder with active manifestations.
* Substance abuse.
* No telephone or means of contacting patient.
* Family household member already enrolled.
* Homeless and not living with relatives/friends.
* Anticipated absence for more than 4 consecutive months.
* Difficulty coming to appointments approximately every 1-2 months
* Already participating in the Diabetes program
* Currently pregnant or intends to get pregnant the next 3 years.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 419 (Actual)
Dates: Start 2003-04; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Framingham Risk Score | 15 months
  Global Cardiovascular disease (CVD) risk score, according to the 1998 sex-specific Framingham point score algorithms of Wilson et al

CONTACTS AND LOCATIONS:
Overall Officials: Randall Stafford, Principal Investigator — Stanford University

REFERENCES:
- [Derived] Ma J, Berra K, Haskell WL, Klieman L, Hyde S, Smith MW, Xiao L, Stafford RS. Case management to reduce risk of cardiovascular disease in a county health care system. Arch Intern Med. 2009 Nov 23;169(21):1988-95. doi: 10.1001/archinternmed.2009.381. PMID 19933961
- [Derived] Berra K, Ma J, Klieman L, Hyde S, Monti V, Guardado A, Rivera S, Stafford RS. Implementing cardiac risk-factor case management: lessons learned in a county health system. Crit Pathw Cardiol. 2007 Dec;6(4):173-9. doi: 10.1097/HPC.0b013e31815b5609. PMID 18091408
- [Derived] Stafford RS, Berra K. Critical factors in case management: practical lessons from a cardiac case management program. Dis Manag. 2007 Aug;10(4):197-207. doi: 10.1089/dis.2007.103624. PMID 17718658